CLINICAL TRIAL: NCT06375668
Title: The Effect of the Probiotic Strains Lactobacillus Plantarum and Lactobacillus Paracasei on Bone Mineral Density in Postmenopausal Women - a Multicenter Randomized Placebo-controlled Study
Brief Title: The Effect of the Probiotic Strains on Bone Mineral Density in Postmenopausal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Biotic Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT/NB/140/2020/PR-MS
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis, Postmenopausal; Bone Density, Low
Keywords: bone mineral density; osteoporosis; probiotics
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Osteoporosis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): A dietary supplement in the form of capsules containing probiotic bacterial strains.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo capsules with the same appearance and weight as probiotic capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The patients who give their consent to take part in this study, will receive one time per day for a period of 12 month a capsule containing ten billions of Lactobacillus plantarum (LP 140 NORDBIOTIC™) and Lactobacillus paracasei (LPC 100 NORDBIOTIC™).
  Arms: Probiotic
Other: Placebo — The patients who give their consent to take part in this study, will receive one time per day for a period of 12 months a capsule containing maltodextrin.
  Arms: Placebo

SUMMARY:
Osteoporosis is a systemic condition characterized by low bone mass and altered bone tissue microarchitecture, with the resulting greater bone fragility leading to fractures. Osteoporosis develops as a result of genetic and environmental factors, with the patient's lifestyle playing an important role. Recent years saw an emergence of reports on the significance of the intestinal microbiota in the development of osteoporosis, thus new ways of modifying the composition and activity of microbiota have been sought, and the potential role of probiotics has been considered. Probiotics are defined as live microorganisms, which-when administered at appropriate doses-are beneficial to the host's health. Probiotics both modify the gut microbiota composition and directly affect the human body. Recently published clinical studies demonstrated that probiotics may facilitate osteoporosis treatment and prevention. The current randomized double-blind placebo-controlled study will assess the effect of a dietary intervention via oral supplementation of Lactobacillus plantarum and Lactobacillus paracasei in a population of Polish postmenopausal women on their bone mineral density assessed via bone densitometry-derived T-scores of the lumbar segment of the spine (L1-L4). Study subjects will take the provided probiotic formulation/placebo orally once daily for 12 months.

DETAILED DESCRIPTION:
The main purpose of the study is to assess the effect of oral probiotic supplementation on bone mineral density in postmenopausal women. A total of 170 female subjects who meet all the inclusion criteria and none of the exclusion criteria are to be included and randomized to one of two arms (the probiotic arm or the placebo arm) at a ratio of 1:1.

The subjects who provide their written informed consent will receive oral probiotic formulation containing a mixture of two strains Lactobacillus plantarum and Lactobacillus paracasei or placebo. The probiotic formulation and placebo will be provided by Nordic Biotic Ltd. (the company will also ensure study drug blinding). Study subjects will take the provided probiotic formulation/placebo orally once daily for 12 months.

The study timeline spans 54 weeks and involves 13 visits, including:

1. Screening visit - subjects eligibility to participate in the study will be assessed based on the inclusion/exclusion criteria - the screening period will last up to 14 before the study drug is administered;
2. Randomization visit (visit 0) - subjects will be randomly allocated to study groups and will receive a supply of the study probiotic or placebo;
3. 6 office visits (at months 2, 4, 6, 8, 10, and 12 of visit 0);
4. 5 remote visits (at months 1, 3, 7, 9, and 11 of visit 0).

All subjects included in the study will undergo:

* History-taking and physical examination at each office visit,
* Nutritional status assessment (measurements of body weight and height, with a BMI calculation) at the screening visit and at months 6 and 12 of the study intervention,
* Two densitometry scans (DEXA) of the lumbar segment of the spine (L1-L4) at the screening visit and at month 12 of visit 0,
* Treatment satisfaction assessment (treatment satisfaction questionnaire) at months 2, 6, 10, and 12 of the study intervention.

At each visit, whether conducted at the doctor's office or remotely, subjects will be asked about their use of the study drug and any gastrointestinal symptoms (number of bowel movements, stool consistency, bloating, abdominal pain), and the use of any other medications (including antibiotics). Each time, the subjects will be also asked about any side effects. Stool consistency will be assessed with the Bristol Stool Form Scale, and abdominal pain, bloating, and nausea will be assessed with a 5-grade Likert scale.

Blood samples will be collected from all subjects during the screening period, after 6 months of intervention and at the completion of intervention (i.e. at month 12).

The following blood tests will be conducted:

1. Complete blood count, erythrocyte sedimentation rate, and C-reactive protein levels (at screening and at months 6 and 12 of the study intervention);
2. Serum calcium, phosphorus, and alkaline phosphatase levels (at screening and at months 6 and 12 of the study intervention);
3. Serum vitamin D and parathormone levels (at screening and at month 12 of intervention).

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women (between 2 and 5 years after their last menstrual period)
2. A dual-energy X-ray absorptiometry (DEXA) scan-based T-score of the lumbar spine (L1-L4) of less than -1.49 (i.e. a normal value according to the World Health Organization)
3. Body mass index (BMI) between 18 and 30
4. Vitamin 25 (OH)D levels between 31-50 ng/mL

Exclusion Criteria:

1. The last menstrual period less than 2 or more than 5 years before study recruitment
2. BMI under 18 or above 30
3. Oral or transdermal hormone therapy with estrogens and/or progestogens within the last 6 months
4. Corticosteroid or thyroid hormone therapy within the last 6 months
5. History of osteopenia or osteoporosis
6. Neoplastic disease treated with cytostatic agents within the last 12 months
7. Autoimmune disorders, including rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis; malabsorption syndromes, including celiac disease; chronic kidney disease; chronic liver failure; endocrine disorders, including Hashimoto thyroiditis, Graves' disease, Cushing disease or syndrome, hyperparathyroidism, hypogonadism, hyperprolactinemia, acromegaly, diabetes mellitus; and other chronic conditions affecting bone metabolism
8. Antibiotic therapy within the last 2 months prior to study recruitment
9. Probiotic use within the last 2 months prior to study recruitment
10. Calcium and vitamin D supplementation within the 2 months prior to study recruitment
11. Treatment with antidepressant or antipsychotic agents involving a change of the agents or dosage within the last 3 months
12. Substance use disorder (alcohol, drugs, nicotine)
13. History of organ transplantation
14. Exposure to the SARS-Cov-2 virus within 14 days prior to study recruitment (based on patient declaration)
15. An acute COVID-19 infection within 14 days prior to study recruitment (based on patient declaration)
16. A surgical procedure scheduled to take place during this study
17. Participation in another study within the last 6 months
18. Inability to give an informed consent in writing
19. Any disease or circumstances that, according to the Investigator or Sponsor, might prevent the subject from completing the study or following study procedures and requirements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
The effect of intervention on bone mineral density | From baseline and after 12 months of intervention
  Bone mineral density (BMD) of the lumbar segment of the spine (L1-L4) will be measured by two densitometry scans (DEXA) and presented as T-score. T-score is measured in standard deviations and reflects the difference between the patient's measured BMD and the mean value of BMD in healthy, young, matched controls (30-year-old women).

SECONDARY OUTCOMES:
Changes in the level of calcium | From baseline and after 6 and 12 months of intervention
  The level of calcium will be measured in serum and expressed in mg/dL.
Changes in the level of phosphorus | From baseline and after 6 and 12 months of intervention
  The level of phosphorus will be measured in serum and expressed in mg/dL.
Changes in the level of alkaline phosphatase | From baseline and after 6 and 12 months of intervention
  The level of alkaline phosphatase will be measured in serum and expressed in U/L.
Changes in the level of vitamin D | From baseline and after 12 months of intervention
  The level of vitamin D will be measured in serum and expressed in ng/mL.
Changes in the level of C-reactive protein | From baseline and after 6 and 12 months of intervention
  The level of C-reactive protein will be measured in serum and expressed in mg/L.
Changes in Body Mass Index (BMI) | From baseline and after 6 and 12 months of intervention
  Weight and height will be combined to report BMI in kg/m2.
Changes in type of stools | From baseline for 12 months of intervention in 1 month intervals
  The stool type will be assessed with the Bristol Stool Formation Scale. The Bristol Stool Formation Scale is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea.
Changes in the number of bowel movements | From baseline for 12 months of intervention in 1 month intervals
  The number of bowel movements per day will be assessed as mean of bowel movements during the last 7 days before visit.
Changes in severity of abdominal pain | From baseline for 12 months of intervention in 1 month intervals
  The severity of pain will be assessed with a patient-defined 5 point Linkert scale: point 0 - no pain, and 1-4 the severity of pain with higher scores indicating worse pain.
Changes in severity of bloating | From baseline for 12 months of intervention in 1 month intervals
  The bloating will be assessed with a patient-defined 5 point Linkert scale: point 0 - no bloating, and 1-4 the severity of bloating with higher scores indicating worse bloating.
Occurrence of adverse events | For 12 months of intervention in 1 month intervals
  Adverse events will be recorded and described throughout the intervention period
Satisfaction with the intervention | At months 2, 6, 10, and 12 of the intervention
  Satisfaction with the intervention will be assessed by a questionnaire consisting of 6 questions regarding satisfaction with the form of the preparation, ease of administration, benefits, and course of treatment on a scale of 1-7, with the higher the score, the higher the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Głogowska-Szeląg, MD, PhD, Principal Investigator — Private Specialist Practice
Locations (3):
- Poland (3):
  - Private Specialist Practice, Bytom
  - Specialist Practice, Katowice
  - Clinical Research Center, Poznan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glogowska-Szelag J, Palka-Kisielowska I, Porawska W, Bierla JB, Szczepankowska AK, Aleksandrzak-Piekarczyk T, Cukrowska B. The Effect of Lacticaseibacillus paracasei LPC100 and Lactiplantibacillus plantarum LP140 on Bone Mineral Density in Postmenopausal Women: A Multicenter, Randomized, Placebo-Controlled Study. J Clin Med. 2024 Oct 8;13(19):5977. doi: 10.3390/jcm13195977. PMID 39408038